CLINICAL TRIAL: NCT02545452
Title: A Parallel Group, Randomized, Open-label Study to Investigate the Effect of the Intravaginally Administered Antimycotic Miconazole, Antibiotic Clindamycin, Spermicide Nonoxynol-9, or Co-usage of Tampons on 3 Consecutive Days on the Pharmacokinetics of Anastrozole and Levonorgestrel Released From an Intra-vaginal Ring in Healthy Young Women
Brief Title: Effect of Concomitant Use of an Antimycotic, an Antibiotic, a Spermicide or Tampons on Pharmacokinetics of Anastrozole and Levonorgestrel Released From Intra-vaginal Ring
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16997; 2014-005167-32 (EudraCT Number)
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Anastrozole; Levonorgestrel; Clotrimazole; Nonoxynol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- BAY98-7196 (Experimental): Investigate the pharmacokinetics effect of a vaginally administered antimycotic (miconazole) during the use of an intra-vaginal ring (IVR) releasing anastrozole (ATZ) and levonorgestrel (LNG)
  Interventions: Drug: Anastrozole / Levonorgestrel (BAY98-7196); Drug: Gyno-Daktarin
- Administered Antibiotic (Experimental): Investigate the pharmacokinetics effect of a vaginally administered antibiotic (clindamycin) during the use of an IVR releasing ATZ and LNG
  Interventions: Drug: Anastrozole / Levonorgestrel (BAY98-7196); Drug: Sobelin vaginal creme
- Administered Spermicide (Experimental): Investigate the pharmacokinetics effect of a vaginally administered spermicide (nonoxynol-9) during the use of an IVR releasing ATZ and LNG
  Interventions: Drug: Anastrozole / Levonorgestrel (BAY98-7196); Drug: Patentex oval
- Tampons (Experimental): Investigate the pharmacokinetics effect of the concomitant use of tampons during the use of an IVR releasing ATZ and LNG; investigate the pharmacokinetics over an extended IVR wearing period of 35 days
  Interventions: Drug: Anastrozole / Levonorgestrel (BAY98-7196); Other: Tampon

INTERVENTIONS:
Drug: Anastrozole / Levonorgestrel (BAY98-7196) — Release rate of the IVR: 1050 μg/d ATZ + 40 μg/d LNG
Drug: Gyno-Daktarin — 400 mg miconazole nitrate per day for 3 consecutive days
  Arms: BAY98-7196
Drug: Sobelin vaginal creme — 100 mg clindamycin 2-dihydrogen phosphat per day for 3 consecutive days
  Arms: Administered Antibiotic
Drug: Patentex oval — 75 mg Nonoxynol-9 per day for 3 consecutive days
  Arms: Administered Spermicide
Other: Tampon
  Other Names: Tampons (3 changes per day) for 3 consecutive days
  Arms: Tampons

SUMMARY:
To investigate the pharmacokinetic effect of a vaginally administered antimycotic (miconazole), antibiotic (clindamycin), spermicide (nonoxynol-9) or the concomitant use of tampons during the use of an intravaginal ring releasing anastrozole and levonorgestrel

ELIGIBILITY:
Inclusion Criteria:

* Healthy pre-menopausal female subject.
* Age: 18 - 50 years (inclusive) at the first screening visit. For the subject > 45 years follicle stimulating hormone (FSH) will be investigated at the second screening visit to confirm the pre-menopausal status (FSH < 40 IU/L in serum).
* Body mass index (BMI ) above or equal 18, and below or equal 30 kg / m² at the first screening visit.
* Adequate venous access.
* Ability to understand and follow study-related instructions
* Agreement to use adequate non-hormonal contraception.
* Confirmation of the subject's health insurance coverage prior to the first screening examination/visit.

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal.
* Thrombophlebitis, venous / arterial thromboembolic diseases (particularly deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction).
* Presence or history of prodromata of thrombosis (e.g. transient ischemic attack, angina pectoris).
* Known hypersensitivity to the study medications (active substances or excipients of the preparations).
* Regular intake of medication other than hormonal contraceptives.
* Use of systemic or topical medication or substances which oppose the study objectives or which might influence them within 4 weeks before first administration of the study medication,
* Smoking of more than 10 cigarettes daily; if the subject is a smoker: subject is older than 35 years
* Suspicion of or known current drug, medicine or alcohol abuse (including anabolics, high-dose vitamins).
* Abnormal cervical smear
* Previous ectopic pregnancy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2016-03-14 (Actual); Study Completion 2016-07-29 (Actual)

PRIMARY OUTCOMES:
Average concentration (Cav) anastrozole after insertion of the intra-vaginal ring for all groups | 202-226h
Average concentration (Cav) anastrozole after insertion of the intra-vaginal ring for all groups | 226-298h
Average concentration (Cav) anastrozole after insertion of the intra-vaginal ring for all groups | 226-384h
Average concentration (Cav) anastrozole after insertion of the intra-vaginal ring for Tampon group | 466-490h
Average concentration (Cav) anastrozole after insertion of the intra-vaginal ring for Tampon group | 490-562h
Average concentration (Cav) anastrozole after insertion of the intra-vaginal ring for Tampon group | 490-648h
Average concentration (Cav) levonorgestrel after insertion of the intra-vaginal ring for all groups | 202-226h
Average concentration (Cav) levonorgestrel after insertion of the intra-vaginal ring for all groups | 226-298h
Average concentration (Cav) levonorgestrel after insertion of the intra-vaginal ring for all groups | 226-384h
Average concentration (Cav) levonorgestrel after insertion of the intra-vaginal ring for Tampon group | 466-490h
Average concentration (Cav) levonorgestrel after insertion of the intra-vaginal ring for Tampon group | 490-562h
Average concentration (Cav) levonorgestrel after insertion of the intra-vaginal ring for Tampon group | 490-648h

SECONDARY OUTCOMES:
Maximum observed plasma concentration before co-medication or tampons (Cmax) | 490h
Time to reach maximum observed concentration before co-medication or tampons (tmax) | 490h
Plasma concentration 28 days after intra-vaginal ring (IVR) insertion (Treatment group D, Day 29) (C(28d)) | 672h
Plasma concentration 35 days after IVR insertion (Treatment group D, Day 36)(C(35d)) | 840h
Average concentration in the extended wearing period (Treatment D, Days 29-36 using the same IVR) | 672-840h
Terminal half-life associated with the terminal slope after removal of IVR (t1/2) | Up to 6 days after IVR removal
Number of participants with adverse events as a measure of safety and tolerability | Up to 14 days after IVR removal

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, Germany